CLINICAL TRIAL: NCT03209284
Title: Influence of the Anatomical Variability of the Maxillary Sinus on New Bone Formation After Transcrestal Augmentation Procedures
Brief Title: Influence of Anatomy of Maxillary Sinus on New Bone Formation After Transcrestal Augmentation Procedures
Acronym: SLSS
Status: Completed | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Collaborators: University of Triste (Unknown)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, DDS, MSc, International Piezosurgery Academy
Other Study IDs: SLSS_IPA
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Atrophy of Edentulous Maxillary Alveolar Ridge
Keywords: maxillary atrophy; transcrestal sinus floor elevation
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bone biopsies were retrieved at the time of implant placement (after 6 months of regenerative procedure) and obtained through implant site preparation with trephine bur
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- narrow sinuses: transcrestal sinus floor elevation in narrow sinuses
  Interventions: Procedure: transcrestal sinus floor elevation
- wide sinuses: transcrestal sinus floor elevation in wide sinuses
  Interventions: Procedure: transcrestal sinus floor elevation

INTERVENTIONS:
Procedure: transcrestal sinus floor elevation — augmentation procedure with xenograft
  Other Names: implant insertion

SUMMARY:
The aim of this study is to analyze neoformed bone after maxillary sinus lifting with transcrestal approach, in atrophic crests (≤5 mm residual bone height). Clinical and laboratory data will be related to maxillo breast anatomy.

DETAILED DESCRIPTION:
Bone resorption and sinus pneumatization, following tooth extraction, are common occurrences in the posterior maxilla. They may cause both a quantitative reduction and qualitative deterioration of bone, resulting in an inadequate bone volume for a standard implant placement. Sinus floor elevation with lateral approach had been described 35 years ago and widely studied afterwards, demonstrating an high predictability in regenerating bone, to allow for reliable implant supported rehabilitations. Maxillary sinus floor elevation with transcrestal approach represents a validated and effective alternative option to vertically enhance the available bone through an access created in the edentulous bone crest. Regardless of graft type, it is not yet well defined how three-dimensional anatomical sinus cavity characteristics may influence healing and mineralization process. An adequate Schneiderian membrane elevation in order to expose sinus floor, buccal and medial walls, seems to represent a crucial factor in influencing new bone formation, as the greatest part of the osteoprogenitor cells derives from these anatomical structures. It is not documented yet the efficacy of the different trnanscrestal sinus floor elevation approaches in exposing the internal bony walls of the sinus. Moreover, on the basis of the fact that only few articles correlated the size of the maxillary sinus with histologic outcome by lateral window and one retrospective radiographic study reported results in relation to the three-dimensional conformation of the sinus using a trans-crestal approach, the investigators conjecture that sinus bucco-palatal diameter could influence the newly-formed bone quality after a crestal sinus lift procedure. For example, the healing in a narrow maxillary sinus could result in a faster new bone formation, when compared to a larger and wider sinus. The aim of this study is to analyze neoformed bone after maxillary sinus lifting with transcrestal approach, in atrophic crests (≤5 mm residual bone height). Clinical and laboratory data will be related to maxillo breast anatomy. The present study has been designed as a multicenter prospective clinical trial. Five clinical centers will treat patients with two-stage transcrestal sinus floor elevation using a calibrated drills technique and a xenogeneic biomaterial. Implants will be inserted 6 months after sinus augmentation and bone-core biopsies will be harvested during the implant site preparation. Histological analyses will be performed in order to assess the quality of the newly-formed tissue and cone beam computed tomography scan examination will be used to evaluate graft resorption over time. For each inserted implant, collection of experimental parameters will be required up to 1 year after its placement.

ELIGIBILITY:
Inclusion Criteria:

Local inclusion criteria will be the following:

* indications for a transcrestal sinus floor augmentation to allow for a single implant placement, based on accurate diagnosis and treatment planning;
* presence of a residual bone crest with a height ≤3 mm on the maxillary sinus in the site where implant placement is programmed;
* the bone crest must be healed (at least three months elapsed after tooth loss);
* age of the patient >18 years;
* patient willing and fully capable to comply with the study protocol;
* written informed consent given.

General exclusion criteria are:

* acute myocardial infarction within the past 2 months;
* uncontrolled coagulation disorders;
* uncontrolled diabetes (HBA1c > 7.5%);
* radiotherapy to the head/neck district within the past 24 months;
* immunocompromised patient (HIV infection or chemotherapy within the past 5 years);
* present or past treatment with intravenous bisphosphonates;
* psychological or psychiatric problems;
* alcohol or drugs abuse.

Exclusion Criteria:

* Local exclusion criterion is the presence of uncontrolled or untreated periodontal disease.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population was composed of all patients presenting for evaluation and management of any partial edentulism requiring unilateral maxillary sinus elevation. To be included in the study sample, patients had to present a residual crestal height on the sinus floor less than 5 mm, to be 18 years or older, and able to understand and sign a written informed consent form.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
newly formed bone | 6 months after surgery
  assessment of newly formed bone via histomorphometric analysis

SECONDARY OUTCOMES:
implant success | 1 years after implant insertion
  short term implant success rate via clinical and radiographic data
exposed walls | 10 day after surgery
  number of sinuses exposed walls after augmentation procedure via cone beam computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr., Principal Investigator — Piezosurgery Academy
Locations (1):
- Piezosurgery Academy, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farina R, Pramstraller M, Franceschetti G, Pramstraller C, Trombelli L. Alveolar ridge dimensions in maxillary posterior sextants: a retrospective comparative study of dentate and edentulous sites using computerized tomography data. Clin Oral Implants Res. 2011 Oct;22(10):1138-1144. doi: 10.1111/j.1600-0501.2010.02087.x. Epub 2011 Feb 15. PMID 21320169
- [Background] Esposito M, Grusovin MG, Rees J, Karasoulos D, Felice P, Alissa R, Worthington H, Coulthard P. Effectiveness of sinus lift procedures for dental implant rehabilitation: a Cochrane systematic review. Eur J Oral Implantol. 2010 Spring;3(1):7-26. PMID 20467595
- [Background] Avila G, Wang HL, Galindo-Moreno P, Misch CE, Bagramian RA, Rudek I, Benavides E, Moreno-Riestra I, Braun T, Neiva R. The influence of the bucco-palatal distance on sinus augmentation outcomes. J Periodontol. 2010 Jul;81(7):1041-50. doi: 10.1902/jop.2010.090686. PMID 20450402
- [Result] Lombardi T, Stacchi C, Berton F, Traini T, Torelli L, Di Lenarda R. Influence of Maxillary Sinus Width on New Bone Formation After Transcrestal Sinus Floor Elevation: A Proof-of-Concept Prospective Cohort Study. Implant Dent. 2017 Apr;26(2):209-216. doi: 10.1097/ID.0000000000000554. PMID 28125520